CLINICAL TRIAL: NCT02399072
Title: A Multicenter, Prospective Epidemiologic Study of the Progression of Geographic Atrophy Secondary to Age-Related Macular Degeneration
Brief Title: A Study of Disease Progression in Participants With Geographic Atrophy Secondary to Age-Related Macular Degeneration
Status: Terminated | Type: Observational
Why Stopped: There is no longer a plan to pursue an approval of lampalizumab.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: GX29639; 2014-003940-11 (EudraCT Number); GX29639 (Other: Hoffmann-La Roche ID)
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geographic Atrophy Participants: Participants with unilateral GA or GA in one eye and choroidal neovascularization (CNV; active or treated) with or without GA, in the contralateral eye, will be evaluated for the progression of GA for up to approximately 60 months.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention administered in this study

SUMMARY:
This study seeks to better characterize relationships between visual function and the progression (worsening) of geographic atrophy (GA) due to age-related macular degeneration (AMD). The study also will generate new information on the relationship between genetics and GA progression. This is a global, prospective, multicenter, epidemiologic study enrolling 200 participants with GA secondary to AMD. The study visits are scheduled to occur every 6 months. The anticipated duration of the study is up to 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Well-demarcated area of GA secondary to AMD
* Women of childbearing potential and men must agree to use adequate contraception for at least 30 days after fluorescein dye administration
* The study is recruiting participants in two different cohorts:

Cohort 1: Participants with unilateral GA OR Cohort 2: Participants with GA in one eye and CNV (active or treated) with or without GA, in the contralateral eye

Exclusion Criteria:

* Previous participation in any studies of investigational drugs for GA / dry AMD (exception for studies of vitamins and minerals)
* GA in either eye due to causes other than AMD
* History of vitrectomy surgery, submacular surgery, or any surgical intervention for AMD
* Previous laser photocoagulation for CNV, diabetic macular edema, retinal vein occlusion, and/or proliferative diabetic retinopathy
* Any ocular/systemic medical conditions that, in the opinion of the investigator, could contribute to participant's inability to participate in the study or interfere with study assessments.
* Requirement for continuous use of therapy indicated in Prohibited Therapy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-08 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline in the GA Area as Assessed by Fundus Autofluorescence (FAF) up to Month 60 | Baseline up to Month 60

SECONDARY OUTCOMES:
Change from Baseline in Best Corrected Visual Acuity (BCVA) Score as Assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) Chart up to Month 60 | Baseline up to Month 60
Change from Baseline in BCVA Score as Assessed by ETDRS Chart Under Low Luminance Conditions up to Month 60 | Baseline up to Month 60
Change from Baseline in Binocular Reading Speed as Assessed by Minnesota Low-Vision Reading Test (MNRead) Cards or Radner Reading Cards up to Month 60 | Baseline up to Month 60
Change from Baseline in Monocular Reading Speed as Assessed by MNRead Cards or Radner Reading Cards up to Month 60 | Baseline up to Month 60
Change from Baseline in Binocular Critical Print Size as Assessed by MNRead Cards or Radner Reading Cards up to Month 60 | Baseline up to Month 60
Change from Baseline in Monocular Critical Print Size as Assessed by MNRead Cards or Radner Reading Cards up to Month 60 | Baseline up to Month 60
Change from Baseline in Near Activity Subscale as Assessed by National Eye Institute Visual Functioning Questionnaire 25-Item Version (NEI VFQ-25) up to Month 60 | Baseline up to Month 60
Change from Baseline in Distance Activity Subscale as Assessed by NEI VFQ-25 up to Month 60 | Baseline up to Month 60
Change from Baseline in Composite Scores as Assessed by NEI VFQ-25 up to Month 60 | Baseline up to Month 60
Change from Baseline in Functional Reading Independence Score up to Month 60 | Baseline up to Month 60
Percentage of Participants With Medical Events | Baseline up to Month 60
Percentage of Participants With Ocular Events | Baseline up to Month 60

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (63):
- United States (11):
  - Retina Specialty Institute, Pensacola, Florida
  - Midwest Vision Research Foundation, Chesterfield, Missouri
  - Char Eye Ear &Throat Assoc, Charlotte, North Carolina
  - Retina Assoc of Cleveland Inc, Cleveland, Ohio
  - Palmetto Retina Center, Florence, South Carolina
  - Tennessee Retina PC., Nashville, Tennessee
  - Retina Res Institute of Texas, Abilene, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - West Virginia University Eye Institute, Morgantown, West Virginia
- Argentina (5):
  - Organizacion Medica de Investigacion, Buenos Aires
  - Oftalmos, Capital Federal
  - Centro Privado de Ojos Romagosa, Córdoba
  - Onnis Instituto oftalmológico privado, Córdoba
  - Oftar, Mendoza
- Australia (4):
  - Marsden Eye Research Centre, Parramatta, New South Wales
  - Adelaide Eye and Retina Centre, Adelaide, South Australia
  - Royal Victorian Eye and Ear Hospital, East Melbourne, Victoria
  - The Lions Eye Institute, Nedlands, Western Australia
- Brazil (2):
  - Instituto da Visão IPEPO, São Paulo, São Paulo
  - Hosp Clinicas da FMUSP, São Paulo, São Paulo
- Canada (6):
  - University of British Columbia, Vancouver, British Columbia
  - QEII - HSC Department of Ophthalmology, Halifax, Nova Scotia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network Toronto Western Hospital, Toronto, Ontario
  - Institut De L'Oeil Des Laurentides, Boisbriand, Quebec
  - Hôpital Maisonneuve - Rosemont, Montreal, Quebec
- France (9):
  - Chi De Creteil; Ophtalmologie, Créteil
  - CHU Bocage; Ophtalmologie, Dijon
  - Hopital de la croix rousse; Ophtalmologie, Lyon
  - Centre Paradis Monticelli; Ophtalmologie, Marseille
  - Centre Odeon; Exploration Ophtalmologique, Paris
  - Hopital Lariboisiere; Ophtalmologie, Paris
  - CHNO des Quinze Vingts; Ophtalmologie, Paris
  - CHU Poitiers - CHR La Miletrie; Ophtalmologie, Poitiers
  - Centres Ophtalmologique St Exupéry; Ophtalmologie, Saint-Cyr-sur-Loire
- Germany (4):
  - Universitäts-Augenklinik Bonn, Bonn
  - Universitätsklinikum Köln; Augenklinik, Cologne
  - Universitätsklinikum Münster; Augenheilkunde, Münster
  - Universitätsklinikum Regensburg, Klinik & Poliklinik für Augenheilkunde, Regensburg
- Hungary (5):
  - Peterfy Sandor utcai Korhaz-Rendelointezet es Baleseti Kozpont, Szemeszet KR, Budapest
  - Semmelweis Egyetem AOK, Szemeszeti Klinika, Budapest
  - Budapest Retina Associates Kft., Budapest
  - Debreceni Egyetem Klinikai Kozpont; Szemeszeti Klinika, Debrecem
  - Ganglion Medial Center, Pécs
- Italy (2):
  - Fondazione Ptv Policlinico Tor Vergata Di Roma;U.O.S.D. Patologie Renitiche, Rome, Lazio
  - ASST FATEBENEFRATELLI SACCO; Oculistica (Sacco), Milan, Lombardy
- Poland (7):
  - OFTALMIKA Sp. z o.o, Bydgoszcz
  - Szpital Specjalistyczny nr 1; Oddzial Okulistyki, Bytom
  - Optimum Profesorskie Centrum Okulistyki, Gdansk
  - Gabinet Okulistyczny Prof Edward Wylegala, Katowice
  - SP ZOZ Szpital Uniwersytecki w Krakowie Oddział Kliniczny Okulistyki i Onkologii Okulistycznej, Krakow
  - Klinika Okulistyczna Jasne Błonia, Lodz
  - SPEKTRUM Osrodek Okulistyki Klinicznej, Wroclaw
- Spain (4):
  - Hospital Universitari de Bellvitge; Servicio de Oftalmologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital General de Catalunya, San Cugat Del Valles, Barcelona
  - Clinica Universitaria de Navarra; Servicio de Oftalmologia, Pamplona, Navarre
  - Institut de la Macula i la retina, Barcelona
- United Kingdom (4):
  - Bradford Royal Infirmary, Bradford
  - Bristol Eye Hospital, Bristol
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - University Hospital Southampton NHS Foundation Trust, Southhampton

REFERENCES:
- [Derived] Salvi A, Cluceru J, Gao SS, Rabe C, Schiffman C, Yang Q, Lee AY, Keane PA, Sadda SR, Holz FG, Ferrara D, Anegondi N. Deep Learning to Predict the Future Growth of Geographic Atrophy from Fundus Autofluorescence. Ophthalmol Sci. 2024 Oct 23;5(2):100635. doi: 10.1016/j.xops.2024.100635. eCollection 2025 Mar-Apr. PMID 39758130
- [Derived] Schmitz-Valckenberg S, Sassmannshausen M, Braun M, Steffen V, Gao SS, Honigberg L, Ferrara D, Pfau M, Holz FG. Interreader Agreement and Longitudinal Progression of Incomplete/Complete Retinal Pigment Epithelium and Outer Retinal Atrophy in Age-Related Macular Degeneration. Ophthalmol Retina. 2023 Dec;7(12):1059-1068. doi: 10.1016/j.oret.2023.07.021. Epub 2023 Jul 29. PMID 37517799
- [Derived] Spaide T, Jiang J, Patil J, Anegondi N, Steffen V, Kawczynski MG, Newton EM, Rabe C, Gao SS, Lee AY, Holz FG, Sadda S, Schmitz-Valckenberg S, Ferrara D. Geographic Atrophy Segmentation Using Multimodal Deep Learning. Transl Vis Sci Technol. 2023 Jul 3;12(7):10. doi: 10.1167/tvst.12.7.10. PMID 37428131